CLINICAL TRIAL: NCT05042739
Title: Early Identification and Predictive Parsing for High Risk Group of Schizophr
Brief Title: Early Identification and Predictive Parsing for High Risk Group of Schizophrenia
Status: Completed | Type: Observational
Sponsor: Wuhan Mental Health Centre (Other)
Collaborators: Health Commission of Hubei Province (Unknown)
Responsible Party: Sponsor
Other Study IDs: ky2018.45
Record Dates: First submitted 2021-08-31; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: High Risk Group of Schizophrenia
Keywords: Psychosis; UHR; CAARMS;SIPS; BSABS
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CAARMS;SIPS; BSABS; — Comprehensive Assessment of At Risk Mental State (CAARMS); Structured Interview for Psychosis-Risk Syndrome (SIPS); Bonn Scale for the Assessment of Basic Symptoms (BSABS);

SUMMARY:
An accurate identification of individuals at ultra-high risk (UHR) based on psychometric tools to prospectively identify psychosis as early as possible is required for indicated preventive intervention. The diagnostic comparability of several psychometric tools is unknown. To address the psychometric comparability of the CAARMS, SIPS and BSABS for subjects who are the immediate family and three-generation blood kinship of patients with schizophrenia. To verify the viability and reliability of the three instruments for these subjects. subjects who all are immediate family and three-generation blood kinship of patients with schizophreniawere interviewed. All the subjects were assessed for a UHR state by three psychometric tools including CAARMS, SIPS and BSABS. The psychometric diagnosis results including at risk of psychosis (UHR+), not at risk of psychosis (UHR-), and Psychosis. Demographic and clinical characteristics interviewed by these three instruments were also measured. The inter-rater agreement was assessed for evaluation of the coherence of the three scales. Transition rates of CAARMS, SIPS and BSABS for UCH+ subjects within 2 years were also recorded.There is good diagnostic agreement between the CAARMS, SIPS and BSABS towards identification of UHR subjects who are immediate family and three-generation blood kinship of patients with schizophrenia. Also, these three instruments are reliable and valid for assessing and detecting at risk mental states in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* all are immediate family and three-generation blood kinship of patients with schizophrenia

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All are immediate family and three-generation blood kinship of patients with schizophrenia diagnosed in Affiliated Wuhan Mental Health Center, Tongji Medical College of Huazhong University of Science & Technology.
  Subjects are recruited from Wuhan Mental Health Center who can be contacted by telephone or an internet homepage.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
The overall agreement percent | 2 years
  diagnostic comparison of CAARMS and SIPS, SIPS and BSABS, CAARMS and BSABS.
the inter-rater reliability | 2 years
  Inter-rater correlation (ICC) coefficients of CAARMS, SIPS and BSABS subscales.
the transition rates of UHR+ to psychosis within 2 years | 2 years
  Transition rates of CAARMS, SIPS and BSABS for UCH+ subjects within 2 years follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, Master, Principal Investigator — Dept. of Psychological Rehabilitation, Affiliated Wuhan Mental Health Center, Tongji Medical College of Huazhong University of Science & Technology
Locations (1):
- Dept. of Psychological Rehabilitation, Affiliated Wuhan Mental Health Center, Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided